CLINICAL TRIAL: NCT04119492
Title: Integrating Brain Imaging and Rehabilitation to Improve Outcomes for Children With Co-occurring DCD & ASD
Brief Title: DCD & ASD Imaging Intervention Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: The Waterloo Foundation (Other)
Responsible Party: Principal Investigator, Jill Zwicker, Principle Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H18-02759
Record Dates: First submitted 2018-12-19; First posted 2019-10-08 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Motor Skills Disorders; Autism Spectrum Disorder
Keywords: developmental coordination disorder; autism; brain imaging; MRI; rehabilitation; CO-OP
MeSH Terms: conditions — Motor Skills Disorders; Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to the CO-OP treatment group or the waitlist control group
Who Masked: Outcomes Assessor
Masking Description: The occupational therapist administering the pre- and post-assessments will be blinded to group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CO-OP Treatment Group (Experimental): Participants in the treatment group will receive occupational therapy once weekly for 10 weeks using the published protocol for the CO-OP approach.
  Interventions: Behavioral: CO-OP Treatment Group
- Waitlist Control Group (No Intervention): Participants in the waitlist control group not receive CO-OP intervention during this time. They will receive their CO-OP intervention 12 weeks after their baseline assessment.

INTERVENTIONS:
Behavioral: CO-OP Treatment Group — Cognitive Orientation to Occupational Performance (CO-OP) is a cognitive approach to solving functional motor problems (Polatajko et al., 2001). Therapists teach children a global problem-solving strategy (Goal-Plan-Do-Check) as means to develop specific strategies for overcoming motor problems; the strategies are determined after a dynamic performance analysis by the therapist to determine where the "breakdown" is in performing the task. Occupational therapists trained in CO-OP will see children for one hour, once weekly for 10 weeks. Parents or caregivers will be encouraged to attend treat¬ment sessions so therapists can instruct them how to facilitate strategy use between treatment sessions. Children will select 3 functional motor goals to be addressed during treatment.
  Arms: CO-OP Treatment Group

SUMMARY:
Developmental Coordination Disorder (DCD) is a neurodevelopmental disorder that affects a child's ability to learn motor skills, such as tying shoelaces, learning to print, or riding a bicycle (APA 2013). It often co-occurs with other conditions, such as Attention Deficit Hyperactivity Disorder (ADHD). Its high co-occurrence with Autism Spectrum Disorder (ASD) has only been permitted since 2013 so it is less well known. Recent neuroimaging studies have begun to unravel the neural underpinnings of each disorder; however, few brain imaging studies have included children with co-occurring DCD and ASD. The first aim of the proposed project is to understand brain structure and function in children with DCD+/-ASD. Despite high co-occurrence of DCD and ASD (Green 2009), motor impairment and functional problems are rarely the focus of therapy for children with ASD. Current best-practice for improving motor function is an approach called Cognitive Orientation to Occupational Performance (CO-OP). The second aim of this study is to examine effectiveness of this treatment approach for children with DCD+ASD and determine if there are brain changes and improvements in motor skills as a result of intervention. This novel project is the first to integrate brain imaging and motor-based rehabilitation in this population and builds on a current study examining brain changes in children with DCD (with and without co-occurring ADHD). Examining the neural basis of these motor difficulties in the presence or absence of co-occurring conditions will help to determine the neural correlates specific to DCD and whether the response to treatment differs in children with co-occurring conditions.

DETAILED DESCRIPTION:
About 5% of children have DCD, a neurodevelopmental disorder that significantly affects their ability to learn motor skills, such as tying shoelaces, learning to print, or riding a bicycle (APA 2013). DCD interferes with school performance, vocational activities, leisure pursuits; it has a lifelong impact, and 75% of children with DCD will continue to experience motor difficulties as adults (Kirby 2014). DCD is highly comorbid with other neurodevelopmental disorders including Autism Spectrum Disorder (ASD) (Green 2009) and Attention Deficit Hyperactivity Disorder (ADHD) (Piek 1999) which exacerbates children's motor and functional problems (Kirby 2014).

Until recently, motor deficits in children with ASD have largely been ignored. Since the Diagnostic and Statistical Manual for Mental Disorders-5th ed. (DSM-5) was published in 2013, a dual diagnosis of ASD and DCD is now permitted. Over 50% of children with ASD have been reported to have DCD (Green 2009), with the degree of motor impairment correlating with autism severity (Dzuik 2007).

The overlap of DCD and ASD is not well-studied, but the high co-occurrence prompts one to wonder whether there are common and distinct neural markers that define these neurodevelopmental disorders. Neuroimaging studies have begun to unravel their neural underpinnings. Abnormalities in the cerebellum (D'Mello 2016; Foster 2015; Liu 2017; Zwicker 2009, 2011) and corpus callosum (Langevin 2014; Frazier 2009) are common to both disorders, but few studies have compared children with DCD and those with co-occurring ASD. Preliminary evidence indicates alterations in network patterns that are unique to the DCD+ASD group when compared to either single diagnosis of DCD or ASD (Caeyenberghs 2016). As one of the first neuroimaging studies to touch upon a dual diagnosis of DCD+ASD, Caeyenberghs et al. found that paralimbic regions exhibit altered connectivity in singular disorders, which are disorder specific to ASD or DCD; however, children meeting criteria for both DCD and ASD exhibit more widespread over-connectivity, specifically in the left association area and medio-occipitotemporal gyrus when compared to DCD alone. While in its infancy, neuroimaging studies suggest that DCD and ASD may have common but also distinct neural underpinnings (Caeyenberghs 2016; Caçola 2017); further research is needed to better understand the neural correlates of each disorder and its co-occurrence.

Current best-practice to improve motor function in children with DCD is Cognitive Orientation to Occupational Performance (CO-OP) (Smits-Engelsman 2013). CO-OP is a task-specific approach designed to improve motor-based skills that a child needs or wants to master; it is a cognitive-based, problem-solving approach that uses verbal mediation and identifies strategies to support skill acquisition (Polatajko 2001). It is largely unknown if children with co-occurring DCD and ASD benefit from CO-OP. Although motor impairment and functional problems are common in ASD, they are rarely the focus of therapy. The primary focus of therapy for children with ASD has always been on social and communication skills or managing sensory processing differences. Preliminary findings from a case study with two children diagnosed with ASD suggest that CO-OP is feasible and able to induce clinically significant improvements in self- and parent-rated performance on each of their motor goals (Rodger 2009). However, a larger sample is needed to confirm these findings.

The CO-OP approach has been effective in meeting child-chosen functional motor goals (Polatajko 2001; Miller 2001), but the neural basis for these improvements is still not known. The investigators are currently investigating brain changes in structure and function associated with CO-OP intervention for children with DCD+/-ADHD and would like to expand their study to include children with co-occurring ASD and DCD. This novel study will help to unravel the brain differences between these co-occurring conditions and explain if and why rehabilitation may benefit children with the dual diagnosis of DCD and ASD.

This study will provide clinicians and researchers with a greater understanding of neurological underpinnings of motor difficulties in children with ASD, and whether interventions should include CO-OP therapy. This project is the first to integrate brain imaging and motor-based intervention in this population and may provide evidence to support new clinical practices to improve outcomes.

RESEARCH DESIGN

Specific Aims and Hypothesis: The proposed study is designed to test the hypotheses that, compared to children with DCD, children with ASD+DCD will exhibit overlapping but distinct differences in brain structure and function, and that rehabilitation associated with brain differences will lead to improvements of motor function. This study builds on the investigators' current CIHR-funded study comparing typically-developing children with children with DCD+/-ADHD and neuroplasticity associated with CO-OP intervention. The proposed study is designed to address the following specific aims:

Aim 1: Characterize brain structure and function in children DCD+ASD and compare results to previously collected data on children with DCD+/-ADHD. Hypotheses: Compared to children with DCD, brains of children with DCD+ASD will show smaller cerebellar volume; differences in microstructural development in motor, sensory, cerebellar, and frontal pathways; and lower correlation between signals from brain regions corresponding to resting-state networks including default-mode, sensorimotor, cerebellar, and frontal networks.

Aim 2: Determine if CO-OP intervention induces neuroplastic changes in brain structure/ function and improves motor skills in children with DCD+ASD. Hypotheses: Compared to a waitlist control group, children in the treatment group will show: (1) strengthened functional connectivity in sensorimotor and cerebellar, and frontal networks; (2) increased integrity of the frontal-cerebellar pathway; (3) increased gray matter volume in the dorsolateral prefrontal, motor, and cerebellar cortices; and (4) improved motor performance. A positive association between functional improvements and changes in brain structure/function is also expected.

Aim 3: Determine if neuroplastic and functional changes are retained at 3-month follow-up. Hypothesis: Children who maintained their functional gains will show increased functional connectivity in brain networks, increased connectivity of the frontal-cerebellar pathway, and increased gray matter volume (as in Aim #2) compared to children who did not maintain their functional gains.

Study Design and Sample Size Calculation: This study is a randomized waitlisted controlled trial. Children will be randomly assigned to either treatment or waitlist group. A statistician will randomize participants using computer-generated sequential blocks of 4 to 6; randomization codes will be kept in sealed opaque envelopes until study enrollment. Added to the investigators' current study, a sample of 30 participants with DCD+ASD will provide > 80% power to detect clinically significant improvement of 2 points on the Canadian Occupational Performance Measure (COPM; Law 2014) [26] (SD of 2.5 and a type-1 error of 0.05) and a 3% difference in axial diffusivity on diffusion tensor imaging, which was correlated with motor function in the investigators' pilot work (Zwicker 2012).

Participants: Thirty children (8-12 years) who meet the diagnostic criteria for DCD and ASD as outlined in the DSM-5 (APA 2013) will be eligible to participate.

Brain Imaging: Prior to MR imaging, children will undergo an MRI simulator session to become familiar with the sights and sounds of the MR environment. All imaging studies will be performed on a state-of-the-art 3-Tesla GE Discovery MR 750 scanner. Brain structure will be assessed using: (1) T1-weighted structural imaging to measure cerebral volume (white matter, cortical gray matter, and deep gray matter) and cerebellar volume, and (2) diffusion tensor imaging (DTI) to measure structural connectivity and white matter microstructure throughout the brain. Brain function will be measured indirectly using resting state MRI to examine functional connectivity at rest in various networks. Total scan time is ~30 min.

Intervention: CO-OP is a cognitive approach to solving functional motor problems (Polatajko 2001). Therapists teach children a global problem-solving strategy (Goal-Plan-Do-Check) as means to develop specific strategies for overcoming motor problems; the strategies are determined after a dynamic performance analysis by the therapist to determine where the "breakdown" is in performing the task. Occupational therapists trained in CO-OP will see children for one hour, once weekly for 10 weeks. Parents or caregivers will be encouraged to attend treatment sessions so therapists can instruct them how to facilitate strategy use between treatment sessions. Children will select 3 functional motor goals to be addressed during treatment, rating their performance and satisfaction of these goals pre- and post-intervention.

Measures: The MABC-2 will be used to assess the degree of motor impairment; scores ≤ 16th percentile indicate DCD (Henderson 2007). This measure provides an overall total score compiled from eight subtests across 3 domains: manual dexterity (3), aiming and catching (2), and balance (3). A commonly used parent questionnaire, the DCDQ (Wilson 2007) will be used to confirm impact of motor skills on daily function. The Conners 3 AI-Parent form will be used to assess ADHD symptomology (Conners 2001). The Social Communication Questionnaire (SCQ), a parent-report questionnaire, will be used to screen for autism-specific social and communication impairments (Rutter 2003).

The primary outcome measure is the COPM (Law 2014), which is an individualized, client-centred measure designed to detect change in a client's self-perception of their performance and satisfaction over time on functional goals that are of importance to them. To supplement the COPM, investigators will video-tape the child performing their 3 motor goals before and after intervention. An occupational therapist blinded to the intervention and pre-test/post-test will score the motor performance using the Performance Quality Rating Scale (PQRS), an objective and observational measure of performance quality (Miller 2001). Fine and gross motor skills will be measured using the short form of the Bruninks-Oseretsky Test of Motor Proficiency 2nd ed. (BOT-2: Bruininks 2005).

Neuroimaging Analysis: DTI: for analyzing diffusion tensor data, tract-based spatial statistics (TBSS) using FMRIB Software Library (FSL) will be conducted. TBSS is a fully automated approach that allows for whole-brain analysis without pre-specification of tracts of interest (Smith 2006). T1-weighted imaging will be analyzed using voxel-based morphometry to compare the local concentration of grey matter between sessions and groups using Statistical Parametric Map-99 package (Ashburner 2000). rs-MRI: FSL will be used to conduct an independent component analysis which allows a data-driven approach to explore resting state networks (Beckman 2005).

Data Analysis:

Aim 1: mean brain volumes will be compared between groups using ANOVAs, with regression-based adjustment for age and sex. Generalized Linear Model will compare DTI measures and functional connectivity timeseries in children with DCD, DCD+ADHD, DCD+ASD, and controls.

Aims 2 & 3: Repeated Measures ANCOVA will be applied to the primary and secondary outcomes to detect changes over time, including effect of maturity in waitlist group, intervention effect in both waitlist and treatment groups, and late effect of intervention in treatment group. Age, MABC-2 scores, and Conners scores will be used as covariates.

ELIGIBILITY:
Inclusion Criteria:

* Children 8-12 years
* Meet the diagnostic criteria for DCD and high-functioning ASD (without intellectual disability) as outlined in the Diagnostic and Statistical Manual - 5th edition
* May have Attention Deficit Hyperactivity Disorder (ADHD) or learning disabilities

Exclusion Criteria:

* Children with metallic objects in their body
* Children with history of claustrophobia

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2019-02-20 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure (COPM) | 12 weeks (before and after intervention)
  Children will rate performance and satisfaction of their three motor goals on a 10-point Likert scale, with higher scores indicating higher performance and satisfaction. A change of 2 points is considered clinically meaningful. The COPM is administered by an occupational therapist not involved in the intervention.
Diffusion Tensor Imaging on MRI | 12 weeks (before and after intervention)
  Fractional anisotropy and diffusivity (mean, axial, and radial)

SECONDARY OUTCOMES:
Performance Quality Rating Scale (PQRS) | 12 weeks (before and after intervention)
  An occupational therapist not involved in the intervention and blinded to pre-test and post-test observes video-recordings of the child performing their three motor goals before and after intervention. The therapist rates the child's movement quality on a scale of 1 to 10, with '1' indicating that the skill is not done at all and '10' indicating that the skill is performed very well. A change of 3-points is considered clinically meaningful.
Bruninks-Oseretsky Test of Motor Proficiency 2nd ed. (BOT-2) short form | 12 weeks (before and after intervention)
  Standardized assessment of motor skills completed by a therapist not involved in the intervention.
Resting-state connectivity on MRI | 12 weeks (before and after intervention)
  Spatial independent components analysis of resting state networks
Voxel-based morphometry | 12 weeks (before and after intervention)
  white matter, cortical gray matter, deep gray matter, and total volumes for cerebrum and cerebellum

CONTACTS AND LOCATIONS:
Overall Officials: Jill G Zwicker, PhD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] American Psychiatric Association, ed. Diagnostic and statistical manual of mental disorders - 5th edition (DSM-5). Washington, DC: American Psychiatric Association; 2013. https://doi.org/10.1176/appi.books.9780890425596.dsm01.
- [Background] Kirby A, Sugden D, Purcell C. Diagnosing developmental coordination disorders. Arch Dis Child. 2014 Mar;99(3):292-6. doi: 10.1136/archdischild-2012-303569. Epub 2013 Nov 19. PMID 24255567
- [Background] Green D, Charman T, Pickles A, Chandler S, Loucas T, Simonoff E, Baird G. Impairment in movement skills of children with autistic spectrum disorders. Dev Med Child Neurol. 2009 Apr;51(4):311-6. doi: 10.1111/j.1469-8749.2008.03242.x. Epub 2008 Feb 3. PMID 19207298
- [Background] Piek JP, Pitcher TM, Hay DA. Motor coordination and kinaesthesis in boys with attention deficit-hyperactivity disorder. Dev Med Child Neurol. 1999 Mar;41(3):159-65. doi: 10.1017/s0012162299000341. PMID 10210248
- [Background] Dziuk MA, Gidley Larson JC, Apostu A, Mahone EM, Denckla MB, Mostofsky SH. Dyspraxia in autism: association with motor, social, and communicative deficits. Dev Med Child Neurol. 2007 Oct;49(10):734-9. doi: 10.1111/j.1469-8749.2007.00734.x. PMID 17880641
- [Background] D'Mello AM, Moore DM, Crocetti D, Mostofsky SH, Stoodley CJ. Cerebellar gray matter differentiates children with early language delay in autism. Autism Res. 2016 Nov;9(11):1191-1204. doi: 10.1002/aur.1622. Epub 2016 Mar 22. PMID 27868392
- [Background] Foster NE, Doyle-Thomas KA, Tryfon A, Ouimet T, Anagnostou E, Evans AC, Zwaigenbaum L, Lerch JP, Lewis JD, Hyde KL; NeuroDevNet ASD imaging group. Structural Gray Matter Differences During Childhood Development in Autism Spectrum Disorder: A Multimetric Approach. Pediatr Neurol. 2015 Oct;53(4):350-9. doi: 10.1016/j.pediatrneurol.2015.06.013. Epub 2015 Jun 25. PMID 26231265
- [Background] Liu J, Yao L, Zhang W, Xiao Y, Liu L, Gao X, Shah C, Li S, Tao B, Gong Q, Lui S. Gray matter abnormalities in pediatric autism spectrum disorder: a meta-analysis with signed differential mapping. Eur Child Adolesc Psychiatry. 2017 Aug;26(8):933-945. doi: 10.1007/s00787-017-0964-4. Epub 2017 Feb 23. PMID 28233073
- [Background] Zwicker JG, Missiuna C, Boyd LA. Neural correlates of developmental coordination disorder: a review of hypotheses. J Child Neurol. 2009 Oct;24(10):1273-81. doi: 10.1177/0883073809333537. Epub 2009 Aug 17. PMID 19687388
- [Background] Zwicker JG, Missiuna C, Harris SR, Boyd LA. Brain activation associated with motor skill practice in children with developmental coordination disorder: an fMRI study. Int J Dev Neurosci. 2011 Apr;29(2):145-52. doi: 10.1016/j.ijdevneu.2010.12.002. Epub 2010 Dec 8. PMID 21145385
- [Background] Langevin LM, Macmaster FP, Crawford S, Lebel C, Dewey D. Common white matter microstructure alterations in pediatric motor and attention disorders. J Pediatr. 2014 May;164(5):1157-1164.e1. doi: 10.1016/j.jpeds.2014.01.018. Epub 2014 Feb 25. PMID 24576693
- [Background] Frazier TW, Hardan AY. A meta-analysis of the corpus callosum in autism. Biol Psychiatry. 2009 Nov 15;66(10):935-41. doi: 10.1016/j.biopsych.2009.07.022. Epub 2009 Sep 12. PMID 19748080
- [Background] Caeyenberghs K, Taymans T, Wilson PH, Vanderstraeten G, Hosseini H, van Waelvelde H. Neural signature of developmental coordination disorder in the structural connectome independent of comorbid autism. Dev Sci. 2016 Jul;19(4):599-612. doi: 10.1111/desc.12424. Epub 2016 May 4. PMID 27147441
- [Background] Cacola P, Miller HL, Ossom Williamson P. Behavioral comparisons in Autism Spectrum Disorder and Developmental Coordination Disorder: A systematic literature review. Res Autism Spectr Disord. 2017 Jun;38:6-18. doi: 10.1016/j.rasd.2017.03.004. Epub 2017 Mar 25. PMID 29057009
- [Background] Smits-Engelsman BC, Blank R, van der Kaay AC, Mosterd-van der Meijs R, Vlugt-van den Brand E, Polatajko HJ, Wilson PH. Efficacy of interventions to improve motor performance in children with developmental coordination disorder: a combined systematic review and meta-analysis. Dev Med Child Neurol. 2013 Mar;55(3):229-37. doi: 10.1111/dmcn.12008. Epub 2012 Oct 29. PMID 23106530
- [Background] Polatajko HJ, Mandich AD, Miller LT, Macnab JJ. Cognitive orientation to daily occupational performance (CO-OP): part II--the evidence. Phys Occup Ther Pediatr. 2001;20(2-3):83-106. PMID 11345514
- [Background] Rodger S, Brandenburg J. Cognitive Orientation to (daily) Occupational Performance (CO-OP) with children with Asperger's syndrome who have motor-based occupational performance goals. Aust Occup Ther J. 2009 Feb;56(1):41-50. doi: 10.1111/j.1440-1630.2008.00739.x. PMID 20854488
- [Background] Miller LT, Polatajko HJ, Missiuna C, Mandich AD, Macnab JJ. A pilot trial of a cognitive treatment for children with developmental coordination disorder. Hum Mov Sci. 2001 Mar;20(1-2):183-210. doi: 10.1016/s0167-9457(01)00034-3. PMID 11471396
- [Background] Law M., Baptiste, S., Carswell, A., McColl, MA., Polatajko, H. & Pollock, N. Canadian Occupational Performance Measure Manual, 5th Edition. Canada. CAOT Publications ACE. 2014.
- [Background] Zwicker JG, Missiuna C, Harris SR, Boyd LA. Developmental coordination disorder: a pilot diffusion tensor imaging study. Pediatr Neurol. 2012 Mar;46(3):162-7. doi: 10.1016/j.pediatrneurol.2011.12.007. PMID 22353291
- [Background] Henderson SE, Sugden DA, Barnett AL. Movement assessment battery for children - 2nd ed. Psychological Corporation London; 2007.
- [Background] Wilson, B.N., Kaplan, B.J., Crawford, S.G., & Roberts, G. (2007). Developmental Coordination Questionnaire 2007 (DCDQ'07). Available at: http://www.dcdq.ca.
- [Background] Conners CK. (2009). Conners3rd Edition (Conners 3). Toronto, ON: Multi-Health Systems.
- [Background] Rutter M, Bailey A. Social communication questionnaire (SCQ). https://www.wpspublish.com/store/p/2954/scq-social-communication-questionnaire. Updated 2003.
- [Background] Bruininks, R., & Bruininks, B. Bruininks-oseretsky test of motor proficiency. 2nd ed. Minneapolis, MN: NCS Pearson; 2005.
- [Background] Smith SM, Jenkinson M, Johansen-Berg H, Rueckert D, Nichols TE, Mackay CE, Watkins KE, Ciccarelli O, Cader MZ, Matthews PM, Behrens TE. Tract-based spatial statistics: voxelwise analysis of multi-subject diffusion data. Neuroimage. 2006 Jul 15;31(4):1487-505. doi: 10.1016/j.neuroimage.2006.02.024. Epub 2006 Apr 19. PMID 16624579
- [Background] Ashburner J, Friston KJ. Voxel-based morphometry--the methods. Neuroimage. 2000 Jun;11(6 Pt 1):805-21. doi: 10.1006/nimg.2000.0582. PMID 10860804
- [Background] Beckmann CF, DeLuca M, Devlin JT, Smith SM. Investigations into resting-state connectivity using independent component analysis. Philos Trans R Soc Lond B Biol Sci. 2005 May 29;360(1457):1001-13. doi: 10.1098/rstb.2005.1634. PMID 16087444
- [Derived] Kangarani-Farahani M, Zwicker JG. White matter changes with rehabilitation in children with Co-occurring autism spectrum disorder and developmental coordination disorder. Neuroimage Rep. 2025 Jun 16;5(3):100272. doi: 10.1016/j.ynirp.2025.100272. eCollection 2025 Sep. PMID 41050947